CLINICAL TRIAL: NCT05956340
Title: Computational Analysis of Spoken Language in Mania
Brief Title: A Study of Spoken Language in Mania
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Mark Frye, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 22-010487
Record Dates: First submitted 2023-07-06; First posted 2023-07-21 (Actual); Last update posted 2025-09-03 (Actual); Status verified 2025-08

CONDITIONS: Manic Episode; Bipolar I Disorder
MeSH Terms: conditions — Mania

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Recording Session During Hospitalization (Experimental): While inpatient, participants will undergo a research interview with recorded audio.
  Interventions: Behavioral: Research interview

INTERVENTIONS:
Behavioral: Research interview — Research interview to capture speech data with high quality cardioid headset microphone

SUMMARY:
This research is being done to find if there are changes with voice and speech during episodes of mania.

ELIGIBILITY:
Inclusion Criteria:

* Provision of informed consent before any study procedures are performed
* English speaker
* Documented clinical diagnosis for Bipolar I Disorder
* Undergoing hospitalization, or boarding in the Emergency Department, for mania as determined by primary clinical staff

Exclusion Criteria:

* Positive urine drug screen for amphetamines or cocaine.
* Expressing paranoid delusions regarding electronic surveillance.
* Documented clinical diagnosis of developmental delay.
* Currently involuntarily hospitalized.
* Deemed at risk for aggression.
* Failure to comprehend study objectives via comprehension questionnaire.
* Individuals who have a guardian and are unable to consent for themselves.
* Current communicable disease requiring isolation.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2023-04-27 (Actual); Primary Completion 2024-09-09 (Actual); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Acoustic Differences | Approximately 48 hours after taking antimanic medications until up to end of subject participation approximately 1 month from enrollment
  The raw audio data will be analyzed for change in pitch, variability of rhythm, and response time.
Syntactical Differences | Approximately 48 hours after taking antimanic medications until up to end of subject participation approximately 1 month from enrollment
  Audio data will be transcribed using voice to text software and then analyzed for syntactical elements of speech including sentence structure and grammar.
Semantic Differences | Approximately 48 hours after taking antimanic medications until up to end of subject participation approximately 1 month from enrollment
  Transcribed audio data will be analyzed for changes in verbosity, lexical diversity, and coherence on a sentence and paragraph level.

CONTACTS AND LOCATIONS:
Overall Officials: Mark Frye, MD, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Minnesota, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials